CLINICAL TRIAL: NCT01640769
Title: MRI Allocation of Pacing Targets in Cardiac Resynchronization Therapy
Brief Title: Imaging Study of Allocation of Pacing Targets in Cardiac Resynchronization Therapy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Libin Cardiovascular Institute of Alberta (Other)
Collaborators: Heart and Stroke Foundation of Canada (Other)
Responsible Party: Principal Investigator, James White, Principal Investigator, University of Calgary
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: MAPIT-CRT
Record Dates: First submitted 2012-07-09; First posted 2012-07-16 (Estimated); Last update posted 2025-06-25 (Actual); Status verified 2025-06

CONDITIONS: Systolic Heart Failure; Dysynchrony; Image Guidance; Digital Twins; Cardiac Resynchronization Therapy
Keywords: Cardiomyopathy; Cardiac Resynchronization Therapy; Image guided therapy; Digital twins; Cardiac Magnetic Resonance Imaging; MRI
MeSH Terms: conditions — Heart Failure, Systolic; Cardiomyopathies

STUDY DESIGN:
Intervention Model Description: 4 dimensional cardiac model to guide optimal delivery of left and right ventricular pacing leads in patients referred for cardiac resynchronization therapy.
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Image guided delivery of pacing leads (Active Comparator): 4D model-guided placement of LV and RV leads to optimal myocardial targets, as derived from pre-procedural Cardiac MRI
  Interventions: Procedure: 4D Model guided delivery of cardiac pacing leads
- Standard delivery of pacing leads (Placebo Comparator): Standard LV and RV lead placement
  Interventions: Procedure: Standard CRT lead delivery

INTERVENTIONS:
Procedure: 4D Model guided delivery of cardiac pacing leads — 4D model-guided placement of LV and RV leads to optimal myocardial targets, as derived from pre-procedural Cardiac MRI
  Arms: Image guided delivery of pacing leads
Procedure: Standard CRT lead delivery — Standard lead delivery
  Arms: Standard delivery of pacing leads

SUMMARY:
This randomized controlled trial will assess a cardiac MRI derived 4D digital cardiac model to optimized left and right ventricular lead delivery to improve response to cardiac resynchronization therapy.

DETAILED DESCRIPTION:
Regional mechanical delay, myocardial scar, and inter-lead distance have each been demonstrated to be relevant variables for the realization of optimal response to cardiac resynchronization therapy (CRT). Pilot study results have suggested clinical feasibility and potential value from LV and RV lead navigation aimed at optimizing these combined variables. A computer software program has been developed to deliver an interactive, 4D digital heart model of mechanical dyssynchrony and myocardial scar to guide LV and RV CRT lead delivery to optimal targets. This multi-center randomized clinical trial has been designed to assess the feasibility, safety and clinical impact of LV-RV lead navigation using a web-deployed 4D cardiac model.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years.
2. Ejection fraction ≤ 35 %.
3. LBBB with QRS duration ≥ 120 msec.
4. NYHA class II-IV.
5. On maximum tolerated heart failure medication therapy ≥ 6 weeks.
6. Clinically accepted for CRT device implantation.

Exclusion Criteria:

1. Failure to provide consent.
2. CCS class III-IV angina.
3. Recent Q-wave myocardial infarction or revascularization procedure ( ≤ 3 months).
4. Atrial fibrillation at time of randomization >6 weeks in duration
5. Standard contra-indications to MRI.
6. Documented severe allergy to intravenous contrast dye ( iodinated CT contrast or Gadolinium MRI contrast).
7. Estimated Glomerular Filtration Rate (eGFR) ≤ 45 ml/min/m2.
8. Patient is pregnant.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 210 (Actual)
Dates: Start 2014-09 (Actual); Primary Completion 2022-01 (Actual); Study Completion 2023-01 (Actual)

PRIMARY OUTCOMES:
Determination of response to image guided placement of cardiac ventricular pacing leads in cardiac resynchronization therapy (CRT) | 6 months
  Cardiac Resynchronization Therapy (CRT) response will be defined as a change in the Left Ventricular Ejection Fraction measured at 6 months post CRT device implant by MUGA (multigated acquisition scan / wall motion study).

SECONDARY OUTCOMES:
All-cause mortality | 12 months
Heart failure hospital admissions | 12 months
improvement in 6-minute hall walk ≥ 30 meters or ≥ 10% | 6 months
  6 minute hallwalk will be done at baseline, 3 months and 6 months
Improvement in New York Heart Association (NYHA) functional class by ≥ 1 | 6 months
  NYHA class will be determined at baseline, 3 months and 6 months (score out of 4)
Improvement in Quality of Life (QOL) score by ≥ 10 points | 6 months
  A "Minnesota Living with Heart Failure" questionnaire will be administered at baseline, 3 months and 6 months (visual analogue score out of 100)
Rate of concordant lead delivery to the "optimal myocardial target" | 6 month
  On the day of procedure, a post lead implant bi-plane fluoroscopy image and PA-LAT CXR will be obtained. These will be reviewed by a core laboratory to score final lead tip (electrode) location using a standardized report form to determine delivery location based on the AHA segmental model.
Total procedural time | 6 month
  Total procedural time from first needle to skin closure, in minutes
Fluoroscopy dose and exposure time | 6 month
  Total fluoroscopy exposure time and radiation dose will be recorded at end of procedure and recorded (in minutes).
Procedural complications | 6 months
  All procedural complications will be recorded following completion of procedure and at 3 and 6 months.
Device complications | 6 months
  All device-related complications, inclusive of need for lead repositioning, will be recorded at 3 months and 6 months.

CONTACTS AND LOCATIONS:
Overall Officials: James White, MD, Principal Investigator — University of Calgary
Locations (5):
- Canada (5):
  - Conect Research, University of Calgary, Calgary, Alberta
  - Halifax Capital Districy Health Authority, Halifax, Nova Scotia
  - Libin Cardiovascular Institute, London, Ontario
  - Ottawa Heart Institute Research Corporation, Ottawa, Ontario
  - University of Laval Research Centre, Québec, Quebec

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Chew DS, Vandenberk B, Exner DV, Labib D, Flewitt J, Mikami Y, Rivest S, Chan D, Manlucu J, Leong-Sit P, Rinne C, Birnie DH, Nery P, Sumner G, Ayala-Paredes F, Philippon F, Yee R, White JA. 4D Digital Heart Model-Guided Left and Right Ventricular Lead Placement for Cardiac Resynchronization Therapy: Results of MAPIT-CRT Trial. Circ Arrhythm Electrophysiol. 2025 Dec 25:e014132. doi: 10.1161/CIRCEP.125.014132. Online ahead of print. PMID 41446931
- [Derived] Laksman Z, Yee R, Stirrat J, Gula LJ, Skanes AC, Leong-Sit P, Manlucu J, McCarty D, Turkistani Y, Scholl D, Rajchl M, Goela A, Islam A, Thompson RT, Drangova M, White JA. Model-based navigation of left and right ventricular leads to optimal targets for cardiac resynchronization therapy: a single-center feasibility study. Circ Arrhythm Electrophysiol. 2014 Dec;7(6):1040-7. doi: 10.1161/CIRCEP.114.001729. Epub 2014 Sep 14. PMID 25221334